CLINICAL TRIAL: NCT02250131
Title: A Multi-center, Randomized Controlled Trial of Goal-directed Perfusion in Cardiac Surgery
Brief Title: The Goal dIrected perFusion Trial in Cardiac Surgery
Acronym: GIFT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director of Cardiothoracic Anesthesia and ICU Dept, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GIFT
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury
Keywords: cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Routine cardiopulmonary bypass technique. Flow adjusted on BSA and temperature
- Goal Directed Perfusion (Active Comparator): Perfusion targeted at oxygen delivery
  Interventions: Procedure: Perfusion targeted at oxygen delivery

INTERVENTIONS:
Procedure: Perfusion targeted at oxygen delivery — Flow on cardiopulmonary bypass based on a target oxygen delivery > 280 mL/min/m2
  Other Names: Cardiopulmonary bypass machine
  Arms: Goal Directed Perfusion

SUMMARY:
Previous studies (1-5) have demonstrated that oxygen delivery (DO2) and carbon dioxide production (VCO2) during cardiopulmonary bypass (CPB) are associated with renal outcome in cardiac surgery. The critical value for DO2 is around 262 - 272 mL/min/m2, and the correspondent critical value of DO2/VCO2 ratio is around 5.0.

Patients with nadir DO2 and DO2/VCO2 ratio below these critical levels have an increased incidence of acute kidney injury (AKI) after cardiac operations.

These observations offer an interpretation for the well-known deleterious effects of excessive hemodilution during CPB, supported by many studies where an association between nadir hematocrit (HCT) on CPB and bad outcomes (especially renal) was found (6-8). It is reasonable to hypothesize that a low oxygen delivery may determine an ischemic damage to the kidney, that due to its peculiar circulation is particularly susceptible to a decrease in the oxygen supply.

However, there is no evidence that a strategy directed towards the specific goal of avoiding critical values of DO2 during CPB may actually decrease the postoperative AKI rate.

The present study is designed to verify the hypothesis that a strategy based on a goal-directed perfusion, aimed to avoid a nadir DO2 below the critical threshold, is effective in limiting the postoperative AKI rate.

DETAILED DESCRIPTION:
2. Study design Multicenter, international, prospective, randomized and controlled study. Patient population

1. Inclusion criteria: Adult (> 18 years) patients undergoing cardiac operations with CPB.

   Expected CPB duration > 90 minutes.
2. Exclusion criteria: severe chronic renal failure (dialysis or serum creatinine > 3.0 mg/dL); emergent (must be operated immediately) procedure; moderate-severe anemia (preoperative HCT < 32%); expected nadir CPB temperature < 32 °C.
3. Withdrawal criteria (after randomization): Need for allogeneic blood transfusions before CPB. Need for allogeneic blood to prime the CPB circuit. DHCA or other violations of the entry criteria. CPB duration below 90 minutes will not be withdrawal criterion, but a subroup analysis is anticipated.

Primary outcomes

Incidence of AKI, defined according to the AKIN criteria (9) as:

AKI stage 1: peak postoperative serum creatinine > 1.5 x baseline or absolute increase 0.3 mg/dL, within the first 48 hours after surgery.

AKI stage 2: peak postoperative serum creatinine > 2.0 x baseline, within the first 48 hours after surgery (AKI stage 3 will be incorporated in the AKI stage 2 group).

Any AKI: stage 1 or higher Peak serum creatinine: within the first 48 postoperative hours. Diagnosis of AKI must be reached within the first 48 hours after surgery, but staging may require a longer time (up to 7 days after surgery).

Secondary outcomes Length of ICU stay (days) Transfusion (red blood cells) rate and amount of red blood cells units transfused Major morbidity (according to STS): mechanical ventilation > 48 hours, AKI stage 2, surgical revision, mediastinitis, stroke.

Operative (in-hospital) mortality 3. Sample size The power analysis is based on the primary outcome "any AKI".

Data from the previous study (1) provide the following figures for the total patient population:

Any AKI rate: 21.2% AKI stage 1: 8.8% AKI stage 2-3: 12.4% With the following distribution according to a cut-off value settled at a nadir DO2 of 280 mL/min/m2.

Outcome All cases N=354 DO2 < 280 mL/min/m2 N= 181 DO2 ≥ 280 mL/min/m2 N= 173 P Any AKI 75 (21.2%) 54 (29.8%) 21 (12.1%) 0.001 AKI stage 1 31 (8.8%) 23 (12.7%) 8 (4.6%) 0.007 AKI stage 2-3 44 (12.4%) 31 (17.1%) 13 (7.5%) 0.006

Based on the above table, we know that the Control Group will spontaneously meet the goal in 50% of the cases, and that will have an any AKI rate of 21%.

We hypothesize that the Goal-Directed Perfusion (GDP) group will meet the goal in 95% of the cases. When the goal is met, the AKIN rate will be 12%; when it is not, it will be 29% This will lead to an expected AKI rate in GDP group of 12.8%.

Therefore, the effect size will be a 40% reduction in the AKI rate (12.8% in GDP group, 21% in Control group.

Based on this effect size, an alpha value of 0.05 and a beta value of 0.20, the number of patients in each group is 350, for a total patient population of 700.

Data analysis will be restricted to patients with a CPB duration > 60 minutes. Same applies to extremely long CPB duration, based on the percentile distribution of CPB.

Interim analyses planned at 25%, 50%, and 75% of patients enrollment, with stopping rules for futility, safety, efficacy. Stopping rule for futility: relative risk for the primary outcome not inclusing the hypothesized value of 0.6 within 99% confidence interval at 50% interim analysis or 95% at 75% interim analysis. Stopping rule for efficacy in presence of a difference in favour of the GDP arm at a P value of 0.01 at 25% interim analysis or 0.05 at the 50% and 75% interim analyses. Stopping rule for safety in presence of a difference in favor of the control arm at a P value of 0.01 at the 25% interim analysis or 0.05 at the 50% and 75% interim analyses (Ethics Committe amendment August 2016).

4. Interventions Patients will be randomly allocated to the Control or the GDP group. Randomization will be performed locally at each participating Institution, using computer-generated schemes.

The patients in control Group will be treated according to the local standards. The patients in GDP group will be treated according to the GDP (see table below).

CONTROL (N=350) TREATMENT (N=350) GDP monitor GDP monitor NO Blood prime (withdrawal) NO Blood prime (withdrawal) Priming volume and nature according to local standards Priming volume and nature according to local standards Perfusion targeted on body surface area and °C Perfusion targeted on DO2 ≥ 280 mL/min/m2 Perfusion pressure according to local standards Perfusion pressure according to local standards Transfusion triggered by HCT according to local standards Transfusion triggered by venous oxygen saturation < 68% and/or oxygen extraction rate > 40% Postoperative care according to local standards Postoperative care according to local standards

Details of the GDP protocol:

The main intervention to achieve the target value of DO2 is increasing the pump flow. Additional interventions include hemofiltration to increase the HCT.

Transfusion protocol

1. During CPB: Transfusions are mandatory below a HCT of 18%. Transfusions are generally prohibited for an HCT > 21%. However, based on the individual judgement that the patient is actually in need for packed red cells, transfusions are allowed between an HCT of 22% and 24%. In this case, this will be considered as a protocol violation, but the patient will not be withdrawn.

   Transfusions are always prohibited for an HCT > 24%.
2. After CPB: HCT < 18%: packed red cells are mandatory HCT between 19% and 23%: packed red cells are allowed HCT between 24% and 30%: packed red cells generally prohibited, but admitted based on physician's judgement. This represents a protocol violation. In this case, this will be considered as a protocol violation, but the patient will not be withdrawn.

HCT > 30%: packed red cells are prohibited.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac operations with CPB. Expected CPB duration > 90 minutes.

Exclusion Criteria:

* Exclusion criteria: severe chronic renal failure (dialysis or serum creatinine > 3.0 mg/dL); emergent (must be operated immediately) procedure; moderate-severe anemia (preoperative HCT < 32%); expected nadir CPB temperature < 32 °C.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative AKI | 48 postoperative hours
  Acute kidney injury defined according to the AKIN criteria (stage 1, stage 2, any AKI, serum creatinine increase)

SECONDARY OUTCOMES:
ICU stay | 15 postoperative days
  lenght of postoperative ICU stay
Transfusion of red blood cells | 15 postoperative days
  Rate of patients receiving red blood cells; amount of red blood cells used
Major morbidity | 15 postoperative days
  Mechanical ventilation > 48 hours, AKI stage 2, surgical revision, mediastinitis, stroke.
Mortality | 30 days after surgery
  Mortality for any cause within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ranucci M. Perioperative renal failure: hypoperfusion during cardiopulmonary bypass? Semin Cardiothorac Vasc Anesth. 2007 Dec;11(4):265-8. doi: 10.1177/1089253207311141. PMID 18270190
- [Result] Ranucci M, Isgro G, Romitti F, Mele S, Biagioli B, Giomarelli P. Anaerobic metabolism during cardiopulmonary bypass: predictive value of carbon dioxide derived parameters. Ann Thorac Surg. 2006 Jun;81(6):2189-95. doi: 10.1016/j.athoracsur.2006.01.025. PMID 16731152
- [Result] Ranucci M, Romitti F, Isgro G, Cotza M, Brozzi S, Boncilli A, Ditta A. Oxygen delivery during cardiopulmonary bypass and acute renal failure after coronary operations. Ann Thorac Surg. 2005 Dec;80(6):2213-20. doi: 10.1016/j.athoracsur.2005.05.069. PMID 16305874
- [Result] de Somer F, Mulholland JW, Bryan MR, Aloisio T, Van Nooten GJ, Ranucci M. O2 delivery and CO2 production during cardiopulmonary bypass as determinants of acute kidney injury: time for a goal-directed perfusion management? Crit Care. 2011 Aug 10;15(4):R192. doi: 10.1186/cc10349. PMID 21831302